CLINICAL TRIAL: NCT05747534
Title: Phase 2a Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Evaluate the Safety and Efficacy of Larazotide (AT1001) for the Treatment of Long COVID in Children and Adults
Brief Title: AT1001 for the Treatment of Long COVID
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boston Children's Hospital, Boston, MA, USA (Other)
Responsible Party: Principal Investigator, Lael Yonker, M.D., Pulmonary Attending Physician, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023P000240
Record Dates: First submitted 2023-02-24; First posted 2023-02-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Long COVID; Long COVID-19; Post Acute COVID-19 Syndrome; Post Acute Sequelae of COVID-19
Keywords: SARS-CoV-2; Long COVID; Pediatrics
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — larazotide acetate

STUDY DESIGN:
Intervention Model Description: Drug arm Placebo arm
  Subjects <25.0 kg will receive 250 µg of AT1001 or placebo, and subjects ≥25.0 kg will receive 500 µg of AT1001 or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind: Participant and Investigator blinded. Pharmacy unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Larazotide Acetate (AT1001) (Experimental): Subjects will receive 250 or 500 µg of Larazotide Acetate orally four times a day (QID) for 21 days. Subjects <25.0 kg will receive 250 µg dose of Larazotide Acetate (AT1001), and subjects ≥25.0 kg will receive 500 µg dose of Larazotide Acetate (AT1001).
  Interventions: Drug: Larazotide Acetate
- Placebo (Placebo Comparator): Subjects will receive 250 or 500 µg of placebo orally four times a day (QID) for 21 days. Subjects <25.0 kg will receive 250 µg dose of placebo and subjects ≥25.0 kg will receive 500 µg dose of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Larazotide Acetate — AT1001 (Larazotide) is a locally acting, non-systemic, octapeptide inhibitor of the zonulin receptor that has shown efficacy in a large variety of animal models of inflammation. The effectiveness of AT1001 in controlling paracellular permeability as a tight junction regulator has been widely demonstrated in animal models both in vitro and in vivo. In MIS-C, prolonged presence of SARS-CoV-2 in the GI tract leads to release of zonulin, a biomarker of intestinal permeability, with subsequent trafficking of SARS-CoV-2 antigens into the bloodstream, leading to hyperinflammation (Yonker, et. al. 2021). Five children treated with AT1001 (through an Emergency Investigational New Drug request authorized by the FDA) displayed a decrease in plasma SARS-CoV-2 Spike antigen levels, inflammatory markers, and symptom improvement superior to that achieved with the current standard of treatment for MIS-C (ie. immunoglobulin, systemic steroids) (Yonker, et. al. 2021) (Yonker, et. al. 2022)
  Other Names: AT1001
  Arms: Larazotide Acetate (AT1001)
Drug: Placebo — Matching placebo will be administered orally four times a day (QID) to participants in the placebo arm.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of Larazotide (AT1001) versus placebo in children and adults 7 to ≤50 years of age who present with symptoms of Long COVID in the presence of SARS-CoV-2 antigenemia. AT1001 (n=100) or placebo (n=50) will be administered orally four times a day (QID) for 21 days.

DETAILED DESCRIPTION:
This is a Phase 2a randomized, double-blind, placebo-controlled clinical trial to evaluate the safety and efficacy of AT1001 for use in children and adults with symptoms of Long COVID. Eligible participants (N= 150) will be treated with AT1001 (n= 100) or matching placebo (n= 50) orally four times a day (QID for 21 days). The study will consist of two phases:

I. Baseline Visit and Treatment phase

After confirming subject eligibility, a licensed physician investigator will obtain informed consent. Subjects will be asked to complete baseline surveys (SBQ™-LC, PedsQL, and Symptom Severity Survey) to assess organ involvement and symptom severity. A venous blood sample will be obtained to, among other things, assess for SARS COV-2 antigenemia (such as Spike protein) and obtain a comprehensive metabolic panel and liver function test. Patients who meet inclusion criteria will be treated with AT1001 or matching placebo at a dose of 250 μg or 500 μg for 21 days. Drug dose will be determined by weight: patients <25.0 kg will receive 250 μg of Larazotide or Placebo, and patients ≥25.0 kg will receive 500 μg of Larazotide or Placebo. Randomization and initial dosing will occur on Visit 1 (Day 1). Visits will then occur on a weekly basis during the treatment phase and will consist of data and/or specimen collection. Visit 2 (Week 1) and Visit 3 (Week 2) will take place virtually and will not involve sample collection. Once the subject has completed 21 days of dosing, Visit 4 (Week 3) will take place in person and require the collection of blood, stool and nasal swabs.

II. Follow-up phase

Patients will have two additional virtual follow-up visits after completing their 21-day course of treatment with the study drug. The first follow up visit will occur one week after completing the study drug (ie. at week 4), and the second will occur one month later (ie. at week 8). Week 8 visit will serve as the end of study visit. Biospecimens will not be collected during the follow-up phase.

Safety monitoring, including physical examination, vitals, and clinical laboratory testing will be performed during the baseline phase and after completion of treatment. Adverse events and concomitant medications will be recorded during the entire study.

Total duration of the participants' participation in the study is approximately 8 weeks (with 21 days treatment period). Total duration of the study is projected to be roughly 42 months, dependent on enrollment timeline.

ELIGIBILITY:
Inclusion Criteria:

* Age 7 to ≤50 years
* History of SARS-CoV-2 infection, documented by positive PCR and/or antigen test
* Ongoing, worsening, new, or recurrent symptoms present ≥4 weeks after SARS-CoV-2 infection.Symptoms include but are not limited to fatigue, malaise, headache, cognitive impairment, neuropsychiatric symptoms, decreased exercise tolerance, post exertional malaise, dyspnea, cough, chest pain, palpitations, tachycardia, gastrointestinal symptoms, musculoskeletal symptoms, fever, lightheadedness, insomnia and other sleep disturbances, anosmia or dysgeusia, pain, paresthesia, menstrual cycle irregularities, erectile dysfunction.

Exclusion Criteria:

* Age ≤6 years or >50 years at time of enrollment
* Pregnancy and/or lactation
* Female participant of childbearing age unwilling to use an acceptable method of birth control for the duration of the study
* Inability to tolerate drug
* Unstable medical conditions or significant co-morbid disease that, by the investigator's determination would make the participant unsuitable for enrollment
* Participation in any other clinical investigation using an experimental drug within 30 days prior to screening
* Intent to participate in another clinical study while participating in this clinical trial
* Blood/plasma donation and or blood loss greater than 400 mL within 90 days, or greater than 200 mL within 30 days prior to screening
* Known hypersensitivity to any of the formulation components of AT1001.
* Abnormal baseline liver function as indicated by AST or ALT ≥3 times the upper limit of normal (ULN), or total bilirubin ≥2x ULN for age
* Abnormal baseline renal function, defined as glomerular filtration rate ≤50 mL/min/1.73m2

Ages: 7 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Event Profiling and Time to Symptom Resolution | 8 weeks
  The primary objective of this study is to evaluate the safety and efficacy of Larazotide (AT1001) versus placebo in children and young adults 7 to ≤50 years of age who present with symptoms of Long COVID. Safety will be assessed by means of adverse event monitoring, and efficacy will be evaluated using the Symptom Burden Questionnaire™ for Long COVID (SBQ™-LC) survey. Additional surveys will be used to monitor symptoms, quality of life and limitation of activities before, during and after treatment with Larazotide or Placebo.

SECONDARY OUTCOMES:
Cytokine profiling, Antigen Testing and Humoral and Cellular Responses | 21 days
  The secondary objective of this study is to characterize the inflammatory response observed in children and young adults 7 to ≤21 years of age with Long COVID and SARS-CoV-2 antigenemia. To assess inflammatory responses, blood, stool and nasal epithelial specimens will be obtained at baseline prior to treatment with Larazotide or Placebo, and at completion of the study's treatment phase (21 days). Inflammatory responses will be evaluated by means of antigen testing, cytokine profiling, among others.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No